CLINICAL TRIAL: NCT00992979
Title: Use of Massage Therapy to Reduce Anxiety and Improve Sleep in Patients Participating in an Inpatient Withdrawal Management (Detox) Program: A Randomized Controlled Pilot Study
Brief Title: Therapeutic Massage to Manage Withdrawal Related Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Holistic Health Research Foundation of Canada (Other)
Responsible Party: Robert William Gilbert, School of Health Sciences, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAL09-01; HHRFC #2007-06
Record Dates: First submitted 2009-10-01; First posted 2009-10-09 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-01

CONDITIONS: Substance Withdrawal Syndrome; Drug Withdrawal Symptoms; Anxiety
Keywords: Addiction; Anxiety; Withdrawal; Psychoactive Drugs; Therapeutic Massage
MeSH Terms: conditions — Substance Withdrawal Syndrome; Anxiety Disorders; Behavior, Addictive | interventions — Massage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Massage (Experimental)
  Interventions: Procedure: Therapeutic Massage
- Relaxation Control (Active Comparator): Relaxation Control Session
  Interventions: Procedure: Relaxation Control

INTERVENTIONS:
Procedure: Therapeutic Massage — Massage therapists with at least 5 years experience will perform the massages. On each of three consecutive days, participants (while fully clothed and in a seated position) will receive a 20-minute back, shoulder, neck and head massage. Subjects will be treated with conventional light pressure Swedish massage techniques which consisted of continuous systematic strokes including kneading and stretching to loosen and rehabilitate the soft tissues of the body and to provide general relaxation. The manual techniques include: effleurage , soothing petrissage , repetitive stroking, rocking , squeezing and mild joint mobilization. As is standard practice in massage therapy delivery, room lights will be dimmed and soft, soothing music played to enhance relaxation during therapy.
  Other Names: Massage
  Arms: Therapeutic Massage
Procedure: Relaxation Control — On each of three consecutive evenings, subjects in this group will participate in a 20 minute relaxation session. This session will be delivered in the same location and with the same lighting and music as with the therapeutic massage group. Each participant will be asked to choose a comfortable position in a chair and a massage therapist will sit quietly in the room approximately 4 feet behind the participant.
  Other Names: Relaxation
  Arms: Relaxation Control

SUMMARY:
In Canada, Addiction Prevention and Treatment Service's (APTS) offer programs specifically designed to help people withdrawal from psychoactive drugs. While participants of withdrawal management (Detox) programs generally reach their goals, the process is a difficult one often exacting an emotional and physical toll. Troublesome symptoms of withdrawal from psychoactive drugs may include anxiety and sleep disturbances. If untreated these symptoms can lead to discontinuation of withdrawal and /or affect the introduction of cognitive-behavioral and or motivational therapy components of Detox programs. In Detox the symptoms of withdraw are managed pharmacologically. Pharmacological tools for managing anxiety and sleep disturbances exist and while effective and safe, in many clinical settings, have limitations and liability in the addiction treatment setting. To address these concerns APTS has incorporated non-pharmacological anxiety management practices into its programs. Prominent among these is therapeutic massage (chair massage in the Swedish tradition). While therapeutic massage has been shown to reduce state and trait anxiety in a variety of clinical settings, no previous study has assessed its anxiolytic or sleep promoting efficacy in an addiction treatment setting. In keeping with ATPS's policy on evidence-based practice, evidence in support of this practice is now required.

Research Objectives: We propose to test the Hypothesis: Therapeutic Massage is an effective therapy for managing withdrawal-related anxiety and for improving sleep effectiveness in patients withdrawing from psychoactive drugs. Our specific objective is to perform a randomized controlled trial (RCT) to determine whether therapeutic massage is effective in comparison to relaxation control treatment in reducing the levels of state and trait anxiety associated with withdrawal and in promoting sleep efficiency.

Research Design: A RCT of the effects of therapeutic massage will be conducted on 80 patients (ages 18-65) attending an APTS Detox program. Patients will be assigned to 1 of 2 treatment groups (n=40/group) and will receive either: therapeutic massage or relaxation control treatment once a day for 3 consecutive days. Anxiety, state and trait, will be measured pre and post each treatment through a standardized tool and physiologic measures (heart rate & blood pre(state and trait) and sleep efficiency will be determined through actigraphy and daily sleep logs.

DETAILED DESCRIPTION:
BACKGROUND Alcohol and Other Drug (AOD) abuse has become a prominent health issue in Canada. According to a recent drug abuse survey, it can be estimated that approximately 2 million Canadians may meet the diagnostic criteria for being dependent upon or having abused AOD. At almost $40 billion/year, the costs of AOD abuse in Canada are substantial. Substance abuse represents a significant drain (both direct and indirect) on Canada's economy, with the largest single direct cost being associated with health care.

The impact on the citizens of Nova Scotia is equally dramatic, as illustrated by the 10,949 individuals who accessed Addiction Services in this province during the 2005 calendar year. 3,252 of these individuals (29.7%) accessed these services through the Addiction Prevention and Treatment Services (APTS), Capital Health. Capital Health exists within the largest integrated academic health district in the Maritimes and provides core health services to 395,000 residents, or 40% of the population of the Nova Scotia and tertiary and quaternary acute care services to residents of Atlantic Canada. Specialized adult health services are provided to a referral population of 550,000 from the rest of the province, as well as to residents of New Brunswick and Prince Edward Island. Of the 3,252 individuals who accessed APTS, Capital Health in 2005, 2020 were male (62.12%) and 1,232 were female (37.88%).

AOD abuse affects people from all walks of life and one prevention and treatment approach cannot be sufficient for all possible forms of abuse. The harms associated with AOD abuse have a significant and detrimental effect on the determinants of health which poses a considerable threat to the social, emotional, physical, and economic well being of Canadian families and communities. Determinants of health are factors impacting on living and working conditions conducive to health in its broadest sense, and include housing, education, genetics, income, employment, culture, physical environment, equity, gender and race. Canada's Drug Strategy (CDS), which was renewed in May 2003, is the federal government's response to addressing the problems associated with the harmful use of AOD, and comprises a series of evidence-based guidelines. Using a comprehensive four-pillar approach, CDS strives to assist individuals, families and communities impacted by substance abuse through education, prevention, harm reduction and enforcement initiatives.

APTS is committed to Canada's Drug Strategy and strives to help individuals, families, and communities of Nova Scotia deal with the harm associated with abuses of AOD. It accomplishes this through a comprehensive range of prevention, intervention and treatment services designed to promote, maintain, and improve health. Included among the services offered by APTS are programs designed to assist in: addiction recovery; withdrawal and management (Detox); tobacco cessation and prevention; substance abuse prevention and community education; women's services; methadone maintenance treatment; and community support groups for gamblers (http://www.cdha.nshealth.ca/programsandservices/addictionprevention/index.html).

The Withdrawal and Management (Detox) program was established at APTS in 1975 and provides care and treatment to approximately 800 individuals each year. This inpatient program consists of detoxification, assessment and education and employs a biopsychosocial approach to treat and empower individuals experiencing the physical/emotional stressors associated with AOD withdrawal. It operates through a supportive community atmosphere that nurtures the difficult process of change. The length of stay in the Detox program depends upon individual assessment, with an average stay of 5 days during which residents participate, under the guidance of nursing staff, in a series of recovery, support and relapse-prevention groups. It is delivered by a staff of 23 full time employees. Detox is available to all individuals residing within the Capital Health district with 15 in-patient beds dedicated to this program. The Detox program integrates a variety of evidence-based pharmacological and biopsychosocial approaches including, but not limited to, behavioral therapy (Wanberg & Milkman, 2002), structured relapse prevention and motivational interviewing (Burke et al., 2003). The participants of the Detox program generally reach their immediate goals, although the process of recovery itself is a difficult one, often exacting an emotional and physical toll. Among the many common and troublesome side effects of the withdrawal process are the development of acute anxiety, sleep disturbances (problems falling asleep or waking frequently) and slight depression (feeling down) which, if left unmanaged, may detrimentally influence the recovery process as well as the ability to engage in further addiction treatment programs.

The need for management of the withdrawal symptoms are quite compelling; lack of sleep exacerbates anxiety and anxiety negatively impacts patient comfort and engagement in working memory tasks (Eysenck, 1985), social interaction (Strahan & Conger, 1998), and prospective memory tasks (Harris & Cumming, 2003). Cumulatively, these negative impacts are of concern in regard to the behavioral therapy attributes of the Detox program. Behavioral therapy is based on the assertion that undesirable behaviors can be replaced by teaching patients new, more desirable ones. It focuses on the patient's responsibility for change and is dependent upon the maintenance of patient comfort and the development of effective, therapeutic relationships (Wanberg & Milkman, 2002). Unchecked anxiety can, and often does, affect the development of these effective relationships. Therefore, the participant may not receive the full benefit of the Detox treatment, potentially leading to decreased overall effectiveness and an increased risk of relapse.

Effective pharmacotherapy's are available for the treatment of anxiety and promotion and maintenance of sleep. Unfortunately, pharmacological therapies are often deemed inappropriate, insufficient or cost-prohibitive in these patient populations. In addressing these concerns, APTS uses a holistic approach to the management of anxiety. While biofeedback techniques and hypnotherapy may be valuable adjuncts for the treatment of anxiety, financial constraints have limited their use at APTS. APTS has chosen to incorporate therapeutic massage and auricular acupuncture into its behavioral therapies, practices that both clinical staff, practitioners and clients report to play an integral role in the success of their addiction recovery program.

Chair massage employing Swedish techniques, currently offered to clients at APTS, consists of continuous systematic strokes including kneading and stretching to loosen and rehabilitate the soft tissues of the body (muscles, tendons and fascia) and to provide general relaxation. The manual techniques include, for example, effleurage (smooth gliding movements intended to evoke the relaxation response), soothing petrissage (lifting, squeezing, wringing, or kneading of soft tissues to increase circulation and to reduce muscle spasm), repetitive stroking (a soothing technique used to decrease sympathetic nervous system firing and to decrease pain perception), rocking (rhythmical side to side motion of a limb or trunk), squeezing (compression of a muscle) and mild joint mobilization (slight distraction and stretch of joint capsules and surrounding tissue). Swedish massage is an inexpensive treatment modality with a low-side effect profile (Ernst, 2003). This treatment has been studied in the management of alcohol withdrawal (Reader et al. 2005), and a recent meta analysis of 37 therapeutic massage studies identified significant reductions in anxiety, blood pressure and heart rate post massage (Moyer et al., 2004). Clinical opinion suggests that the most profound benefits accrue to those most in need, e.g. individuals experiencing physical or emotional stressors (Rattray & Ludwig, 2000).

RATIONALE For the vast majority of clinical disciplines, the delivery of therapy is defined by a series of highly structured treatment regimes. In contrast, the delivery of care for the treatment of addiction is far less structured. This reflects the fact that unlike most other clinical conditions, the manifestations of addiction are highly variable, both at the level of patients and communities. As such, the service delivery framework provided by individual addiction treatment centers possess varying degrees of distinctness, with each centre granted the freedom to apply combinations of biopsychosocial approaches that they believe best suits their specific patient population. Health Canada now recommends the application of evidence-based decision making principles in all areas of research and clinical practice. The implementation of evidence-based principles has lead clinicians and researchers alike to identify a variety of challenges in addiction treatment programs in Canada. Included among these is an absence of defined behavioral outcomes or evidence of efficacy for many of the programs offered. Even more surprising is the realization that some long entrenched therapies have never been empirically verified for their general efficacy or the subpopulations which they might best serve (e.g. alcohol, drugs, gambling and/or combinations there in). Given the impact that addiction has on the social and economic fabric of Nova Scotia, many in the addiction treatment field are now asking the question "How effective is our particular addiction treatment program and can it be improved?" Today therapeutic massage is used in addiction treatment programs across North America and Europe and was first initiated as an outreach program to APTS by the Canadian College of Massage and Hydrotherapy in 2005. Among experienced clinical professionals, the belief is strong that therapeutic massage plays an important role in managing the level of anxiety in their patients. However, no peer-reviewed scientific study has ever been performed to test the efficacy of therapeutic chair massage in reducing acute anxiety and improving sleep quality in patients participating in an addiction recovery setting. This is of importance in light of the fact that Health Canada now recommends the use evidence-based decision making principles in all areas of research and clinical practice.

STATEMENT OF RESEARCH QUESTION One area in need of attention at APTS is our use of complementary and alternative therapies like therapeutic chair massage and auricular acupuncture. While numerous studies have illustrated the effectiveness of therapeutic massage in reducing anxiety (Moyer et al., 2004), no experimental study has been designed to test its anxiolytic or sleep enhancement effects in an addiction treatment setting. Today we are challenged with the task of substantiating the efficacy of this apparently important component of our addiction treatment program.

The objective of this application is test the HYPOTHESIS: Therapeutic massage (chair massage utilizing Swedish techniques) is an effective therapy for the management of acute recovery-related anxiety and for promoting sleep onset and improved sleep efficiency in patients attending the Detox program at APTS.

Our Specific Objective is:

a) To perform a randomized controlled trial to determine whether therapeutic massage is effective, compared with relaxation control treatment, in reducing the level of state and trait recovery-related anxiety and in promoting sleep onset and improved sleep efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Individuals receiving inpatient treatment for withdrawal from psychoactive drugs and who were able to give informed consent and comply with study procedures were eligible to participate.
* being at least 18 years of age;
* self-reported primary presenting problem as one of the following: alcohol, cocaine, or opioids

Exclusion Criteria:

* prior treatment or experience with massage therapy
* prior history of anxiety or sleep disorder
* history of coagulation or platelet disorders or be currently taking medications that may promote bleeding
* contraindications to the treatment intervention as described in the standards of care of the College of Massage Therapists of Ontario (http://www.cmto.com/regulations/standard.htm).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety (Spielberger State Trait Anxiety Inventory of Adults (Y1 and Y2)) | State and trait anxiety scores will be determined at baseline (at the time of recruitment into the study) and then immediately prior to and within 10 minutes following each intervention session (pre/post design)

SECONDARY OUTCOMES:
Heart Rate and Blood Pressure | Heart rate and blood pressure will be measured at baseline (at the time of recruitment into the study) and then immediately prior to and within 10 minutes following each intervention session (pre/post design)
Sleep Quality | On each intervention day subjects will wear an actigraph during normal sleep time. They will also be asked to complete a sleep log in the morning, upon waking for each post-intervention day

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Gilbert, PhD, Principal Investigator — Dalhousie University; Shaun Black, MSc, Study Director — Capital District Health Authority, Addiction Prevention and Treatment Services; Kathleen Jacques, PhD, RMT, Study Director — Canadian College of Massage and Hydrotherapy
Locations (1):
- Addiction Prevention and Treatment Services; Capital District, Halifax, Nova Scotia, Canada